CLINICAL TRIAL: NCT04033094
Title: Baseline Epidemiologic Assessment of Abuse-Deterrence of MorphaBond ER (BEAD-MB) (PMR 2961-9)
Brief Title: Baseline Epidemiologic Assessment of Abuse-Deterrence of MorphaBond Extended Release (BEAD-MB)
Acronym: BEAD-MB
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: MORPH-A-U403
Record Dates: First submitted 2019-07-18; First posted 2019-07-25 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Baseline Epidemiologic Assessment
Keywords: Abuse; Misuse; Overdose
MeSH Terms: conditions — Drug Overdose | interventions — Morphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MorphaBond ER
  Interventions: Drug: MorphaBond ER
- Comparator Group
  Interventions: Drug: Comparator Drug

INTERVENTIONS:
Drug: MorphaBond ER — This was a retrospective, non-interventional study. Previous users of branded and generic products (tablets or capsules) with ER and immediate release (IR) release type formulations of oxycodone, oxymorphone, hydromorphone and morphine (except MorphaBond).
  Groups: MorphaBond ER
Drug: Comparator Drug — This was a retrospective, non-interventional study. Previous users of the MorphaBond ER brand of ER morphine sulfate with A-D labeling, by prescription or non-prescription.
  Groups: Comparator Group

SUMMARY:
The main objectives of this study are to provide surveillance/descriptive data to (a) assess utilization of MorphaBond ER and selected comparators overall and by age group and census regions using nationally-projected quarterly drug dispensing data and (b) assess the scope and pattern of abuse and clinical outcomes for MorphaBond ER using nationally representative data or data from large geographic areas in different populations.

Findings of this study will support the design of formal epidemiology assessment of the risks of addiction, overdose, and death outcomes associated with MorphaBond ER and appropriate comparators in the future.

DETAILED DESCRIPTION:
The study started after the launch of MorphaBond ER in October 2017 and will continue until September 2020 and the final study report will be submitted to the FDA by December 2020.

This is an observational study that will provide descriptive data on the utilization and abuse of MorphaBond ER and related outcomes (addiction, misuse, abuse, overdose, overdose-related deaths) for MorphaBond ER and selected comparators in response to the US-FDA's post-marketing requirement (PMR 2961-9 for MorphaBond ER).

No investigational products or pharmaceutical agents will be provided or administered for the purpose of this study. Multiple data sources, representing different populations and large geographic areas in the US, will be utilized to study the patterns of MorphaBond ER utilization and abuse and related outcomes.

The overall purpose of this study is to collect meaningful baseline data to support subsequent studies for formal epidemiologic assessment of abuse deterrence of MorphaBond ER as required by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* MorphaBond ER users or relevant comparator users

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MorphaBond ER users and relevant comparator users
Sampling Method: Non-Probability Sample
Enrollment: 17566 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Quarterly number of MorphaBond Extended Release (ER) dosage unit dispensed | October 2017 through September 2020
Percentage and rates of abuse/abuse-related outcomes of MorphaBond Extended Release (ER) vs. comparators | October 2017 through September 2020
Rates of misuse of MorphaBond Extended Release (ER) vs. comparators | October 2017 through September 2020
Rates of addiction of MorphaBond Extended Release (ER) vs. comparators | October 2017 through September 2020
Overdose rates of MorphaBond Extended Release (ER) vs. comparators | October 2017 through September 2020
Overall mortality rates and opioid overdose death rates of MorphaBond Extended Release (ER) vs. comparators | October 2017 through September 2020

SECONDARY OUTCOMES:
Number and proportion of abuse-related outcomes by routes of administration (e.g. ingestion, inhalation, etc). | October 2017 through September 2020

CONTACTS AND LOCATIONS:
Overall Officials: Safety Study Director, Study Director — Daiichi Sankyo
Locations (1):
- Daiichi Sankyo, Inc., Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No